CLINICAL TRIAL: NCT02351882
Title: Safety and Efficacy of Nabilone in Alzheimer's Disease: a Pilot Study
Brief Title: Safety and Efficacy of Nabilone in Alzheimer's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 318-2013
Record Dates: First submitted 2014-11-17; First posted 2015-01-30 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer Disease; Agitation; Weight Loss; Pain; Oxidative Stress
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Weight Loss; Pain | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nabilone (Active Comparator): Participants randomized into the nabilone arm will be prescribed nabilone for 6 weeks. After one-week placebo washout, they will be taking placebo for an additional 6 weeks.
  Interventions: Drug: Nabilone
- Placebo (Placebo Comparator): Participants randomized into the placebo arm will be receiving placebo for 6 weeks. After one-week placebo washout, they will be prescribed nabilone for an additional 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Participants randomized to nabilone treatment arm, will undergo a one-week placebo washout, followed by 6 weeks of nabilone treatment (weeks 1-6). Participants will then receive a one-week placebo washout (week 7), before receiving 6 weeks of placebo treatment (weeks 8-14).
  Arms: Nabilone
Drug: Placebo — Participants randomized to placebo arm, will undergo a one-week placebo washout, followed by 6 weeks of drug matched placebo (weeks 1-6). Participants will then receive a one-week placebo washout (week 7), before receiving 6 weeks of nabilone treatment (weeks 8-14).
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is commonly associated with behavioural changes such as agitation. Severe agitation is important to treat because it not only increases progression of AD and physical health problems (increased falls and weight loss), but it also decreases quality of life and increases caregiver stress. Currently prescribed treatments (i.e., antipsychotics) for agitation in AD do not work in everybody and when they do work the effect is small and they increase the risk of harmful side effects, including death. As a result, there is an urgent need for safer medication options. The cannabinoid nabilone can now be prescribed in capsule form for appetite and pain killing effects. Nabilone's calming effects may benefit those with agitation, and help the weight loss and untreated pain frequently associated with agitation. Through a clinical trial, the investigators hope identify the benefits of nabilone in the treatment of agitation in AD.

The investigators objective is to determine whether nabilone is an efficacious and safe treatment for agitation, as well as having benefits for pain, weight and behavioural symptoms. This will be a 14 week clinical trial (participants take nabilone for 6 weeks, placebo for 6 weeks (order randomized) with 1 week between treatments). The investigators will assess and compare agitation, weight, pain, memory, behaviour and safety.

Nabilone is a new class of medication that may be a safe and effective treatment for agitation in AD, with added benefits on appetite and pain. Reducing these symptoms would increase quality-of-life and reduce caregiver stress.

DETAILED DESCRIPTION:
Objectives: The investigators objective is to provide pilot data addressing whether the ∆9-tetrahydrocannabinol (THC) analogue nabilone is a pharmacological option for managing agitation, a particularly difficult to treat neuropsychiatric symptom (NPS), as well as having benefits for pain, weight and overall NPS, and gather double-blind information on tolerability and safety. This group of symptoms is particularly prevalent in patients with moderate to severe AD.

Rationale: The high prevalence and impact of agitation in patients with moderate to severe Alzheimer's disease (AD) makes this neuropsychiatric symptom (NPS) a key determinant of decreased quality of life. Associated with agitation are weight loss, and pain, both of which lead to additional loss of quality of life. Agitation frequently necessitates use of antipsychotics, which, while well-studied, have modest efficacy and severe side effects including increased mortality. With the development of synthetic THC analogues, the therapeutic potential of cannabinoids can now be evaluated. Cannabinoids can be prescribed as capsules to treat anorexia and pain in certain patient groups. In addition to these potentially beneficial effects on appetite and pain, a recent study suggested positive effects of nabilone on agitation in dementia. Importantly, in addition to psychotropic effects, emerging evidence suggests neuroprotective (inhibit Aβ-induced microglial activation and excitotoxicity) and anti-inflammatory abilities, which can decrease oxidative stress, in stark contrast to the negative effects of antipsychotics. As such, this system is of high potential relevance in agitated patients with AD.

Research Plan: This will be a randomized cross-over study comparing 6 weeks of nabilone and placebo, with a 1 week placebo washout preceding each treatment phase in Long-term care (LTC) patients, and outpatients with moderate to severe AD and agitation. Study outcomes will be measured at baseline and end of treatment for each treatment phase. The primary outcome measure will be the Cohen-Mansfield Agitation Inventory (CMAI). The secondary outcomes will be the weight (kg), overall NPS (Neuropsychiatric Inventory (NPI)), NPI agitation/aggression subscale, nutrition (Mini Nutritional Assessment - Short Form (MNA-SF), body mass index (BMI), skin fold thickness), pain (The Pain Assessment In Advanced Dementia (PAINAD)), cognition (Mini-Mental State Examination (MMSE); Severe Impairment Battery (SIB)) and clinical significance (Alzheimer's Cooperative Study-Clinician Global Impression of change (ADCS-CGIC). Safety (heart rate, blood pressure, and adverse events) will also be assessed at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥55 years of age
* Diagnostic and Statistical Manual (DSM) -V criteria for Major Neurocognitive Disorder due to AD. Patients with both Major Neurocognitive Disorder due to AD and Major Vascular Neurocognitive Disorder (i.e., mixed AD and cerebrovascular disease) will also be included.
* Currently in moderate-to-severe stage of dementia (Mini-Mental Status Examination (MMSE) ≤24)
* Presence of clinically significant agitation (Neuropsychiatric Inventory (NPI) agitation subscale ≥3)
* If treated with cognitive-enhancing medications (cholinesterase inhibitors and/or memantine), dosage must be stable for at least 3 months. If the ChEI and/or memantine has been discontinued, they may enroll after 1 month.

Exclusion Criteria:

* Change in psychotropic medications less than 1 month prior to study randomization (e.g., concomitant antidepressants)
* Contraindications to nabilone (history of hypersensitivity to any cannabinoid)
* Current or past significant cardiovascular disease (e.g. uncontrolled hypertension, ischemic heart disease, arrhythmia and severe heart failure)
* Presence or history of other psychiatric disorders or neurological conditions (e.g. psychotic disorders, schizophrenia, stroke, epilepsy), previous or current abuse of/dependence on marijuana

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in agitation; Cohen-Mansfield Agitation Inventory (CMAI) | baseline (0 weeks) to 14 weeks
  A 29-point scale that measures agitation in two dimensions, verbal and physical, each of which having two poles, aggressive and non-aggressive.

SECONDARY OUTCOMES:
Change in neuropsychiatric symptoms; Neuropsychiatric Inventory (NPI) | baseline (0 weeks) to 14 weeks
  A widely used assessment of behaviour disturbances in dementia, including: apathy, agitation, delusions, hallucinations, depression, euphoria, aberrant motor behaviour, irritability, disinhibition, anxiety, sleeping, and eating. The frequency and severity of these symptoms are judged on a 4-point and 3-point scale, respectively. A 5-point scale is used to evaluate caregiver distress.
Change in cognition; Standardized Mini-mental State Examination (sMMSE) | baseline (0 weeks) to 14 weeks
  Used to describe cognitive impairment.
Change in cognition; Severe Impairment Battery (SIB) | baseline (0 weeks) to 14 weeks
  Used to describe cognitive impairment for severe AD.
Change in cognition; Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) | baseline (0 weeks) to 14 weeks
  Used to describe cognitive impairment for moderate AD.
Change in clinical representation; Alzheimer's Disease Cooperative Study - The Clinician Global Impression (ADCS - CGIC) | 2 to 14 weeks
  The ADCS-CGIC is used to measure overall clinically significant change in patients.

OTHER OUTCOMES:
Change in pain; Pain Assessment In Advanced Dementia (PAINAD) | baseline (0 weeks) to 14 weeks
  The PAINAD is a 5-item observer-rated scale conducted after a 5-minute observation. The scale examines breathing, vocalizations, facial expression, body language, and consolability.
Change in nutritional status; Mini Nutritional Assessment - Short Form (MNA-SF) | baseline (0 weeks) to 14 weeks
  The MNA-SF is a structured interview consisting of 6 items that categorizes patients as malnourished, at risk of malnutrition, or of normal nutritional status.
Change in heart rate | baseline (0 weeks) to 14 weeks
  Heart rate will be assessed at weeks 0 to 14 to monitor safety.
Change in levels of blood biomarkers | baseline (0 weeks) to 14 weeks
  Biomarkers will be obtained from blood work.
Change in blood pressure | baseline (0 weeks) to 14 weeks
  Blood pressure will be assessed at weeks 0 to 14 weeks to monitor safety.

CONTACTS AND LOCATIONS:
Overall Officials: Krista L. Lanctôt, PhD, Principal Investigator — Sunnybrook Research Institute; Nathan Herrmann, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ruthirakuhan MT, Herrmann N, Gallagher D, Andreazza AC, Kiss A, Verhoeff NPLG, Black SE, Lanctot KL. Investigating the safety and efficacy of nabilone for the treatment of agitation in patients with moderate-to-severe Alzheimer's disease: Study protocol for a cross-over randomized controlled trial. Contemp Clin Trials Commun. 2019 May 23;15:100385. doi: 10.1016/j.conctc.2019.100385. eCollection 2019 Sep. PMID 31338476
- [Result] Herrmann N, Ruthirakuhan M, Gallagher D, Verhoeff NPLG, Kiss A, Black SE, Lanctot KL. Randomized Placebo-Controlled Trial of Nabilone for Agitation in Alzheimer's Disease. Am J Geriatr Psychiatry. 2019 Nov;27(11):1161-1173. doi: 10.1016/j.jagp.2019.05.002. Epub 2019 May 8. PMID 31182351
- [Result] Ruthirakuhan M, Herrmann N, Andreazza AC, Verhoeff NPLG, Gallagher D, Black SE, Kiss A, Lanctot KL. 24S-Hydroxycholesterol Is Associated with Agitation Severity in Patients with Moderate-to-Severe Alzheimer's Disease: Analyses from a Clinical Trial with Nabilone. J Alzheimers Dis. 2019;71(1):21-31. doi: 10.3233/JAD-190202. PMID 31322567
- [Result] Ruthirakuhan M, Herrmann N, Andreazza AC, Verhoeff NPLG, Gallagher D, Black SE, Kiss A, Lanctot KL. Agitation, Oxidative Stress, and Cytokines in Alzheimer Disease: Biomarker Analyses From a Clinical Trial With Nabilone for Agitation. J Geriatr Psychiatry Neurol. 2020 Jul;33(4):175-184. doi: 10.1177/0891988719874118. Epub 2019 Sep 23. PMID 31547752
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852
- [Derived] Ruthirakuhan M, Lanctot KL, Vieira D, Herrmann N. Natural and Synthetic Cannabinoids for Agitation and Aggression in Alzheimer's Disease: A Meta-Analysis. J Clin Psychiatry. 2019 Jan 29;80(2):18r12617. doi: 10.4088/JCP.18r12617. PMID 30753761